CLINICAL TRIAL: NCT04655235
Title: Translational Investigation of the Glutamatergic and GABAergic System in Schizophrenia - a Combined EEG-, FMRI-, Genetic, Serological and Cell Biological Study
Brief Title: Translational Investigation of the Glutamatergic and GABAergic System in Schizophrenia
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Arnim Gaebler, Jun.-Prof. Dr. med. Arnim Johannes Gaebler, RWTH Aachen University
Other Study IDs: 19-201
Record Dates: First submitted 2020-11-28; First posted 2020-12-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First visit: 10 mL EDTA-blood for genetic analysis and 20 mL blood for serological analysis Second visit: 20 mL EDTA-blood for reprogramming of iPSC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- patients with schizophrenia: 200 patients with a DSM 5- diagnosis of schizophrenia
  Interventions: Genetic: Genotyping
- healthy relatives of patients with schizophrenia: 200 healthy relatives of the patients with schizophrenia
  Interventions: Genetic: Genotyping
- healthy control subjects: healthy control subjects without relatives with mental disorders
  Interventions: Genetic: Genotyping

INTERVENTIONS:
Genetic: Genotyping — Genotyping of glutamatergic, GABAergic, dopaminergic and other CNS-related genes

SUMMARY:
In the last years, the imbalance between excitatory and inhibitory neuronal activity has come to the fore as a possible molecular disease mechanism of schizophrenia . Pharmacological studies have suggested different fMRI and EEG markers of that molecular dysfunction (resting state connectivity changes, auditory mismatch and steady state deficits). However, previous research is inconclusive regarding their genetic basis, their reliability, inter-individual relationship as well as disease specificity. Therefore, in this study we aim at estimating the effect sizes, test-retest-reliability and clinical correlates of the respective markers in a comparative fashion in patients with schizophrenia, their relatives and healthy control subject. To assess their molecular validity, we will assess their relationship with glutamatergic and GABAergic genotypes and cellular disease models. The proof of such a relation would give the opportunity of detecting a glutamatergic and GABAergic imbalance throughout non-invasive imaging. Furthermore, it would help deepening our understanding of the molecular pathophysiology of mental disorders which will be essential for the development of more effective drugs.

DETAILED DESCRIPTION:
The participant collective will include 3 groups of 200 persons, consisting of patients with schizophrenia, their healthy relatives and healthy controls that are not related to the patients. The patients must be diagnosed of schizophrenia according to DSM-5 to be included in the study and will be excluded when there is a further psychiatric comorbidity that dominates in the clinical appearance. All participants have to be aged from 18 to 80 years, be mentally and contractually capable to give their consent to study participation and may not be pregnant or have a structural neurological disease. The healthy participants must not suffer from a psychiatric disorder themselves and, additionally, the control subjects must not have psychiatric disorders in the family history of their first-degree relatives.

Every participant will undergo the same examinations, tests and measurements. All subjects will be taken a blood sample of 30 milliliters of blood that will be tested for antibodies against the NMDA receptor, neuronal growth factors, components of the glutamatergic and GABAergic metabolism and markers for the integrity of the blood brain barrier. In addition to that, a genetic analysis to identify risk alleles for schizophrenia and important glutamatergic and GABAergic genes will be performed. A medical history of every subject will be taken, including medication, somatic and psychiatric disorders. Furthermore, a row of psychiatric ratings scales as well as neuropsychological and neurological tests will be performed.

These will include

* Structured Clinical Interview for DSM Disorders (SCID)
* Mini-RDoC
* Short Form Health 36 (SF-36)
* Personal and Social Performance Scale (PSP)
* Positive and Negative Syndrome Scale
* Berner Psychopathologie-Skala
* Calgary Depression Rating Scale for Schizophrenia
* Conners' Adult ADHD Rating Scales (CAARS)
* Wender Utah Rating Scale (WURS-k)
* Clinical Global Impression (CGI)
* Global Assessment of Functioning (GAF)
* Extrapyramidal Symptom Rating Scale (EPS)
* Heidelberg Neurological Soft Signs Scale
* Brief Assessment of Cognition in Schizophrenia
* d2 test

Every study participant must undergo an EEG measurement while different, neutral visual (fixation cross or movies without sound) and auditive stimuli (tones or clic trains) will be presented to them. They will be instructed to ignore the auditive stimuli. Resting state, auditory steady state response (ASSR) and two different auditory mismatch paradigms will be used. Without contradiction for the conduction of an MRI measurement, a combined EEG/ MRI measurement and a pure MRI measurement (without EEG) using the same paradigms are intended. It will also include structural (T1, T2 and diffusion tensor imaging) MRI and MR spectroscopy of glutamate and GABA. All the previously mentioned examinations are planned to take place on the same day with an approximate expenditure of time of five hours. If necessary, the examinations may also take place on different days, providing that there will be a maximum of three weeks between the first and the last measurement. Except from the blood withdrawal, we intend repeating all the measurements for a second time. This repetition must take place at least one day and not later than three years after the first measurement. It will not be necessary to repeat the clinical and neuropsychological tests if the first testing does not date back more than 6 weeks. In a second part of the study, we want to generate induced pluripotent stem cells (iPS cells) from 15 participants of every study group. For this purpose, a further blood sample of 20 milliliters of blood must be taken. The participants of the second part of the study will be selected based on special genetic, EEG or fMRI characteristics revealed in the first part of the study if they agree to be contacted again.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* diagnosis of schizophrenia according to DSM-5
* aged 18 to 80
* being mentally and contractually capable to give their consent to study participation

Exclusion Criteria:

* pregnancy
* structural neurological disease
* a further psychiatric comorbidity that dominates in the clinical appearance

HEALTHY PARTICIPANTS

Inclusion Criteria:

* aged 18 to 80
* being mentally and contractually capable to give their consent to study participation

Exclusion Criteria:

* pregnancy
* structural neurological disease
* psychiatric disorder
* for healthy controls: psychiatric disorders in the family history of first-degree relatives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from the Department of Psychiatry, Psychotherapy and Psychosomatics at Uniklinik RWTH Aachen, Alexianer Krankenhaus and the psychiatric institutions of Katharina Kasper ViaNobis GmbH in Gangelt.
  The patients will be asked whether their healthy relatives may be contacted in terms of study participation. Additionally, they will be handed the study teams' contact details. Relatives suffering from the same psychiatric disorder as the patients can also be included and will be contacted the same way as the healthy relatives.
  Healthy controls will be searched via notices in the Uniklinik RWTH Aachen.
  Furthermore, we will contact former study participants that have given their consent to being contacted for a renewed study participation.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
MMN | 1 day to maximum 3 years
  Mismatch negativity amplitude
ASSR Power | 1 day to maximum 3 years
  40-Hz auditory steady state response spectral power

SECONDARY OUTCOMES:
ASSR Phase Locking | 1 day to maximum 3 years
  40-Hz auditory steady state response phase locking
Functional connectivity | 1 day to maximum 3 years
  Whole brain resting state functional connectivity matrix
Psychopathology as assessed with the PANSS | 1 day to maximum 3 years
  Positive and negative syndrome scale (Minimum: 30, Maximum: 210, higher scores mean worse outcome)
Psychopathology as assessed with the BPP | 1 day to maximum 3 years
  Berner Psychopathologie-Skala (Minimum: -3, Maximum: +3, higher positive scores mean excessive speech, movements or higher positive affect, higher negative scores mean a lack of speech, movements or higher negative affect,
Psychopathology as assessed with the CGI | 1 day to maximum 3 years
  Clinical Global Impression (CGI) (Minimum: 1, Maximum: 7, higher scores mean worse outcome)
Electrophysiology | one appointment of additional blood sampling to isolate cells for iPSC reprogramming
  Electrophysiology assessed in iPSC derived neurons obtained from subsamples using patch clamp and microelectrode array recordings
Expression of neural markers in iPSC derived neurons | one appointment of additional blood sampling to isolate cells for iPSC reprogramming
  quantitative polymerase chain reaction (qPCR), immunofluorescence, western blot
Neurological status as assessed with the EPS | 1 day to maximum 3 years
  Extrapyramidal Symptom Rating Scale (Minimum: 0, Maximum: 4, higher scores mean worse outcome)
Neurological soft signs assessed with the Heidelberg Scale | 1 day to maximum 3 years
  Heidelberg Neurological Soft Signs Scale (Minimum: 0, Maximum: 75, higher scores mean worse outcome)
Psychopathology as assessed with the SCID | 1 day to maximum 3 years
  Structured Clinical Interview for DSM Disorders (SCID)
Psychopathology as assessed with the Mini-RDoC | 1 day to maximum 3 years
  Minimum data set Research Domain Criteria
Psychopathology as assessed with the SF-36 | 1 day to maximum 3 years
  Short Form Health (Minimum: 0, Maximum: 100, higher scores mean better outcome)
Psychopathology as assessed with the PSP | 1 day to maximum 3 years
  Personal and Social Performance Scale (Minimum: 1, Maximum: 100, higher scores mean better outcome)
Psychopathology as assessed with the CDSS | 1 day to maximum 3 years
  Calgary Depression Rating Scale for Schizophrenia (Minimum: 0, Maximum: 27, higher scores mean worse outcome)
Psychopathology as assessed with the CAARS (Minimum: 0, Maximum: 198, higher scores mean worse outcome) | 1 day to maximum 3 years
  Conners' Adult ADHD Rating Scales
Psychopathology as assessed with the WURS-k (Minimum: 0, Maximum: 84, higher scores mean worse outcome) | 1 day to maximum 3 years
  Wender Utah Rating Scale
Psychopathology as assessed with the GAF | 1 day to maximum 3 years
  Global Assessment of Functioning
Neuropsychology assessed with BACS | 1 day to maximum 3 years
  Brief Assessment of Cognition in Schizophrenia
Neuropsychology assessed with d2 test | 1 day to maximum 3 years
  d2 test

CONTACTS AND LOCATIONS:
Overall Officials: Arnim Gaebler, M.D., Principal Investigator — Uniklinik RWTH Aachen
Locations (3):
- Germany (3):
  - Alexianer Hospital, Aachen, Northrine-Westphalia
  - ViaNobis - Die Fachklinik, Gangelt, Northrine-Westphalia
  - University hospital RWTH Aachen, Aachen

IPD SHARING:
Plan to Share IPD: No